CLINICAL TRIAL: NCT06794619
Title: Clinical Study to Assess the Effects of Prebiotic and Probiotic Supplement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Olly, PBC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: OLLCLI1F
Record Dates: First submitted 2025-01-06; First posted 2025-01-27 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Healthy
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Oral dietary supplement. Instructions: Take 1 gummy per day with or without food or water. Do not take more than 1 gummy per day.
  Interventions: Dietary Supplement: Placebo
- Dietary Supplement with actives (Active Comparator): Oral dietary supplement. Instructions: Instructions: Take 1 gummy per day with or without food or water. Do not take more than 1 gummy per day.
  Interventions: Dietary Supplement: Dietary Supplement with actives

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo
  Arms: Placebo
Dietary Supplement: Dietary Supplement with actives — Dietary Supplement containing probiotic and prebiotic ingredients
  Arms: Dietary Supplement with actives

SUMMARY:
Randomized, Crossover, Double-Blind, Placebo-Controlled, Single-Center Clinical Study with Daily Food Log, Stool Samples, Blood Draws, and Validated Questionnaires (GSRS, Bristol stool chart, and DQLQ) with Oral Dietary Supplement

ELIGIBILITY:
Inclusion Criteria:

* Subject is a healthy male or female between the ages of 18 - 50 years, inclusive;
* Subject indicates they have mild or moderate occasional digestive issues (bloating or mild discomfort) with no diagnosed chronic digestive or immune conditions;
* Subject has signed a written Informed Consent and is willing and able to attend all visits and comply with study instructions;
* Subject agrees to maintain their regular diet and exercise habits;
* Subject agrees to limit alcohol consumption to 1 drink per day or no more than 7 drinks per week.
* Females Only: Female subject of childbearing potential must agree to be on a form of birth control for at least 6 months prior to screening visit. Acceptable forms of birth control are: Abstinence (not having heterosexual sex), same-sex partner, double barrier (condom, diaphragm, or cervical cap with spermicidal foam, gel, or cream), vasectomized partner for at least 6 months prior to the screening visit. Birth control (such as the pills, intravaginal ring, or the arm implant) are not acceptable forms of birth control.
* Subject agrees not to take any dietary supplements or medications throughout the clinical study;
* Subject agrees to have four blood draws taken at the testing facility and agrees to collect stool samples (four times) as instructed.
* Subject has an active email address and is capable of completing online questionnaires.

Exclusion Criteria:

* Subject has severe digestive issues (e.g., IBS, Crohn's Disease, Ulcers, Severe Constipation, etc.);
* Subject has allergies to dietary supplements or their ingredients;
* Subject is currently taking medication(s) for a chronic condition;
* (Females of Child Bearing Potential only) Subject is pregnant, nursing, or planning to become pregnant;
* Subject has significant past/current medical history (e.g., previous diagnosis of gastrointestinal or metabolic conditions, cancer, liver or kidney disease);
* Subject has any disease or condition (e.g., hepatic, multiple sclerosis, high blood pressure, renal, Thrombosis/Phlebitis, cardiac, pulmonary, digestive, hematological, neurological, locomotor or psychiatric disease) which in the opinion of the Investigator would compromise the safety of the subject;
* Subject has travel plans and would be unable to attend all study visits;
* Subject is currently taking any dietary supplements, vitamins and/or medications;
* Subject is currently taking probiotics related to digestion or any products that may impact gut microbiota (e.g. probiotic supplements, yogurt, and/or fermented drinks);
* Subject has used antibiotics in the last 3 months;
* Subject has a positive medical history for cancer within the past 5 years;
* Subjects has any planned surgeries and/or invasive medical procedures during the study;
* Subjects is considered unreliable or unlikely to be available for the duration of the study;
* Subject is an employee of the clinical site or the sponsor

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Changes in Gastrointestinal Symptoms (GSRS) Scores | from enrollment to end of study at 10 weeks
  Weekly GSRS scores will be analyzed to assess changes in the severity and frequency of gastrointestinal symptoms across the active and placebo arms.
  Data will be compared between the active supplement and placebo groups and within each participant across different time points to measure crossover effects.
Changes in Stool Consistency (Bristol Stool Chart) | from enrollment to end of study at 10 weeks
  Daily stool consistency ratings will provide data on changes in bowel health and regularity.
  Average stool consistency scores will be compared across baseline, active treatment, and placebo phases.

SECONDARY OUTCOMES:
Changes in Immune Biomarkers (Blood Samples) Levels | from enrollment to end of study at 10 weeks
  Blood sample analysis will focus on immune function biomarkers counts. Changes in immune biomarkers will be compared between baseline, active treatment, and placebo periods.
Changes in Gut Microbiome Composition (Stool Samples) | from enrollment to end of study at 10 weeks
  Stool samples will be analyzed for changes in microbial diversity and specific bacterial populations, which may indicate changes in gut health.
  Comparisons will be made between active treatment and placebo periods to identify any significant shifts in the microbiome.

OTHER OUTCOMES:
Changes in Daily Quality of Life (DQLQ) Scores | from enrollment to end of study at 10 weeks
  DQLQ scores will be compared across different phases to assess any impacts of the supplement on participants' well-being and daily functioning.
  Changes in quality of life will be analyzed at baseline, end of each treatment period, and post-washout.
Changes in Daily Diet and Symptoms (Daily Diary) | from enrollment to end of study at 10 weeks
  Changes in daily food intake, symptom levels, and stool consistency from the diaries will be analyzed to identify any patterns or correlations between dietary habits and digestive health outcomes. This data will provide exploratory insights into lifestyle factors that may influence supplement effects.
Changes During Initial Dose Effects (24-Hour Questionnaire) | from enrollment to end of study at 10 weeks
  Short-Term Effects on Symptoms (24-Hour Data). The 24-hour questionnaire data following the initial dose will be used to capture any immediate digestive effects of the supplement.
  Changes in reported symptoms within this initial period will be compared between the active supplement and placebo groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Princeton Consumer Research, St. Petersburg, Florida, United States